CLINICAL TRIAL: NCT02701036
Title: Sporadic Degenerative Ataxia With Adult Onset: Natural History Study (SPORTAX-NHS)
Brief Title: Sporadic Degenerative Ataxia With Adult Onset: Natural History Study
Acronym: SPORTAX-NHS
Status: Recruiting | Type: Observational
Sponsor: Ataxia Study Group (Other)
Collaborators: German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Klockgether, Prof. Dr. Thomas Klockgether, Ataxia Study Group
Other Study IDs: SPORTAX 010/05
Record Dates: First submitted 2016-01-28; First posted 2016-03-08 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Late Onset Sporadic Cerebellar Ataxia
Keywords: sporadic ataxia; MSAc; SAOA; multiple system atrophy of cerebellar type; natural history

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — 2x9 ml EDTA blood samples. Blood samples are taken according to established protocols for future genetic studies. The samples are sent to the Department of Medical Genetics (Tübingen, Germany).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- sporadic adult onset ataxia: SAOA denotes the non-hereditary degenerative adult-onset ataxia disorders that are distinct from multiple system atrophy (MSA). SAOA is a group of ataxia of unknown etiology characterized by a slowly progressive cerebellar syndrome starting around the age of 50 years. Possibly is accompanied by signs of mild autonomic dysfunction that do not meet the criteria of severe autonomic failure required for a diagnosis of MSA.
- cerebellar multiple system atrophy: Multiple system atrophy of cerebellar type is a cerebellar syndrome with sporadic onset developing in midlife, with autonomic features of otherwise unexplained bladder dysfunction with or without erectile dysfunction in males, orthostatic hypotension and atrophy of the cerebellum, brainstem, and middle cerebellar peduncles.

SUMMARY:
The key goals of SPORTAX-NHS is to compare the phenotype of multiple system atrophy of cerebellar type (MSA-C) and sporadic adult onset ataxia of unknown aetiology (SAOA) and to determine the rate of disease progression in both groups including determination of the factors that predict the development of MSA-C vs. SAOA, and at which time after onset of ataxia, a reliable distinction between both disorders is possible.

The planned study will also allow to collect blood samples and other biomaterials from patients with sporadic ataxia, which will be useful for future genetic and biomarker studies.

DETAILED DESCRIPTION:
Progressive ataxia frequently starts in adults without a familial background. These patients may suffer from an acquired ataxia or a genetically determined ataxia despite negative family history. In the majority of them, however, a genetic or acquired cause of ataxia cannot be identified suggesting a sporadic degenerative ataxia. They can be subdivided into two groups. In one group, the underlying brain disease is multiple system atrophy (MSA), specifically MSA of cerebellar type (MSA-C). The characteristic clinical feature of MSA is the presence of severe autonomic failure defined by orthostatic hypotension or urinary incontinence. The second group is distinguished from MSA-C by the lasting absence of severe autonomic failure. These patients have been designated as sporadic adult onset ataxia of unknown aetiology (SAOA). In the first years after ataxia onset, a distinction between MSA-C and SAOA is often not possible.

There are only few studies comparing the phenotype of MSA-C and SAOA, and longitudinal studies focussing on the evolution of the phenotype of these disorders are completely lacking. In particular, the progression rate of SAOA compared to MSA-C has not been defined. In addition, it is unknown which factors predict the development of MSA-C vs. SAOA, and at which time after onset of ataxia, a reliable distinction between both disorders is possible.

To answer these questions, we plan to create a European registry of patients with sporadic degenerative ataxia of adult onset and to perform a natural history study. The planned study will also allow to collect blood samples and other biomaterials from patients with sporadic ataxia, which will be useful for future genetic and biomarker studies.

ELIGIBILITY:
Inclusion Criteria:

* Progressive ataxia
* Disease onset after the age of 40 years
* Informative and negative family history (no similar disorders in first- and second-degree relatives; parents older than 50 years, or, if not alive, age at death of more than 50 years, no consanguinity of parents)

Exclusion Criteria:

* No established acquired cause of ataxia

Clinical exclusion criteria:

* No onset of ataxia in association with stroke, encephalitis, sepsis, hyperthermia or heat stroke;
* no chronic diarrhea;
* no unexplained visual loss;
* no alcohol abuse;
* no chronic intake of anticonvulsant drugs;
* no other toxic causes; no malignancies;
* no rapid progression (development of severe ataxia in less than 12 weeks);
* no insulin-dependent diabetes mellitus

Imaging exclusion criteria:

* No evidence of multiple sclerosis, ischemia, hemorrhage or tumor of the posterior fossa;
* absence of signal abnormalities on T2/FLAIR-images except abnormalities compatible with MSA

Laboratory exclusion criteria:

* Negative molecular genetic testing for FRDA (only required if there is no cerebellar atrophy on MRI, SCA1, SCA2, SCA3, SCA6, FMR1 premutation (only required if prominent tremor, cognitive impairment and signal abnormality on T2/FLAIR images in the middle cerebellar peduncle);
* antineuronal antibodies negative (only required, if disease duration less than 3 years);
* normal levels of vitamin B12;
* VDRL negative;
* normal thyreoid function

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with adult onset degenerative ataxia, in which acquired and genetic causes of ataxia have been excluded.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-04; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Scale for the assessment and rating of ataxia (SARA) | through study completion, an average of 10 years
  Both conditions (SAOA and MSAc) are part of neurodegenerative diseases, chronic progressive disorders. Their disease progression, can be measured using a validated ataxia scale, SARA. SARA was evaluated in two large validation trials performed by the EUROSCA clinical group and was found to be easy to use, reliable, and valid.

SECONDARY OUTCOMES:
Inventory of non-ataxia signs (INAS) | through study completion, an average of 10 years
  The occurrence of accompanying non-ataxia symptoms is recorded using INAS.
spinocerebellar ataxia functional index (SCAFI) | through study completion, an average of 10 years
  to assess the severity of ataxia in an objective way, three quantitative tests, 8m-walk, 9HPT (hole peg test) and PATA rate (timed speech task) are used.
Unified Multiple System Atrophy Rating Scale (UMSARS) | through study completion, an average of 10 years
  UMSARS is a validated scale for multiple system atrophy used to assess additional symptoms typically occurring in MSA. The scale comprises the following components: Part I, historical, 12 items; Part II, motor examination, 14 items; Part III, autonomic examination; and Part IV, global disability scale.
Questionnaire for Cerebellar Multisystem Atrophy diagnostic criteria | through study completion, an average of 10 years
  To distinguish between SAOA and MSAc adjusted criteria for multiple system atrophy of cerebellar type on the basis of consensus statement on the diagnostic criteria for MSAc are used (Second consensus statement on the diagnosis of multiple system atrophy: Neurology. 2008 Aug 26; 71(9): 670-676).
  Probable MSAc requires a sporadic, progressive adult-onset disorder including rigorously defined autonomic failure and cerebellar ataxia. Possible cerebellar MSA requires a sporadic, progressive adult-onset disease including cerebellar ataxia and at least one feature suggesting autonomic dysfunction plus one other feature that may be a clinical or a neuroimaging abnormality (Babinski sign with hyperreflexia, Stridor, Parkinsonism (bradykinesia and rigidity), Atrophy on MRI of putamen, middle cerebellar peduncle, or pons, Hypometabolism on FDG-PET in putamen, Presynaptic nigrostriatal dopaminergic denervation on SPECT or PET. If both criteria are not met patient is classified as a SAOA.
EQ-5D | through study completion, an average of 10 years
  Health related Quality of life is assessed using EQ-5D, a generic instrument that has been developed and validated by the EuroQuol Group (1990) and is available in validated translations for use as a questionnaire.
PHQ-9 | through study completion, an average of 10 years
  Assessment of depressive symptoms is done using a validated 9-item short form of the Patient Health Questionnaire (PHQ), a questionnaire that has been developed to screen for psychiatric co-morbidity in unselected populations
Comparison of phenotype of cerebellar multiple system atrophy and sporadic adult onset ataxia of unknown etiology | through study completion, an average of 10 years
  classified as "SAOA" can convert into MSAc, that is why they are followed with yearly clinical assessments.
RBDSQ | through study completion, an average of 10 years
  REM Behaviour Disorder Screening Questionnaire (RBDSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klockgether, MD, Principal Investigator — Department of Neurology, Bonn, Germany
Locations (14):
- Department of Neurology, Medical University, Innsbruck, Innsbruck, Austria
- Germany (9):
  - Universitätsmedizin Berlin Charité, Berlin
  - Department of Neurology, University of Bonn, Bonn
  - Department of Neurology, University Clinic Essen, University of Duisburg-Essen, Essen
  - Department of Neurology, University of Frankfurt, Frankfurt
  - Hamburg UKE Abt. Neuropädiatrie, Hamburg
  - Otto-von-Guericke Universität Magdeburg, Magdeburg
  - Friedrich-Baur-Institut an der Neurologischen Klinik, München
  - Universitätsmedidzin Rostock - Klinik und Poliklinik für Neurologie, Rostock
  - Dept. of Neurodegenerative Diseases Tübingen, Tübingen
- Italy (2):
  - Department of Neuroscience, Federico II University Naples, Naples
  - Universita cattolica del sacro cuore, Rome
- Radboud University Medical Center, Department of Neurology, Donders Institute for Brain, Cognition, and Behaviour, Nijmegen, Netherlands
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Giordano I, Harmuth F, Jacobi H, Paap B, Vielhaber S, Machts J, Schols L, Synofzik M, Sturm M, Tallaksen C, Wedding IM, Boesch S, Eigentler A, van de Warrenburg B, van Gaalen J, Kamm C, Dudesek A, Kang JS, Timmann D, Silvestri G, Masciullo M, Klopstock T, Neuhofer C, Ganos C, Filla A, Bauer P, Tezenas du Montcel S, Klockgether T. Clinical and genetic characteristics of sporadic adult-onset degenerative ataxia. Neurology. 2017 Sep 5;89(10):1043-1049. doi: 10.1212/WNL.0000000000004311. Epub 2017 Aug 9. PMID 28794257
- See also: Sportax Database — http://www.ataxia-study-group.net/html/studies/sportax